CLINICAL TRIAL: NCT03582800
Title: Subcutaneous Injection of Sodium Thiosulfate for Ectopic Calcifications or Ossifications. A Pilot Study
Acronym: ITS-PILOT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I17004 (ITS-PILOT)
Record Dates: First submitted 2018-06-13; First posted 2018-07-11 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Systemic Sclerosis; Dermatomyositis; iPPSD2
Keywords: Sodium thiosulfate; Ectopic calcification; Ectopic Ossification
MeSH Terms: conditions — Scleroderma, Systemic; Dermatomyositis; Ossification, Heterotopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treated (Experimental): M0-M6: run-in phase (control) M6-M12: STS treatment phase
  Interventions: Drug: STS

INTERVENTIONS:
Drug: STS — M0-M6 (run-in phase): medical care and follow-up as usual
  M6-M12 (STS phase):
  * Patients with iPPSD2 will be treated with subcutaneous infusion using a portable pump.
  * Patients with dermatomyositis or systemic sclerosis will be treated with repeated injections every two weeks.
  Patients will receive a maximal total number of 11 STS injections. M12: final visit (V5): clinical evaluation, photograph and CT scan of the treated lesion, pain and quality of life evaluation.

SUMMARY:
Ectopic soft tissue calcifications or ossifications can complicate the course of numerous diseases; most of them are rare or very rare. Even if the clinical, radiological and pathological presentation of ectopic calcifications and ossifications are different, the same hypotheses are discussed considering their hypothetical pathophysiology. Indeed, high calcium phosphate product, local cellular lesions and abnormal transdifferentiation of mesenchymal cells are regularly evoked when pathophysiology of such calcifications or ossifications are discussed. Apart from several case reports that have not been confirmed so far, no medical treatments are available, leading to significant pain and impairment of quality of life for patients. Therefore, only surgical treatment can be proposed when the volume or the consequences of these calcifications/ossifications become too important.

Sodium thiosulfate (STS) is currently used as a cyanide poisoning antagonist and a chemoprotectant against adverse effects of several chemotherapies such as Cisplatin. Numerous case reports and several studies have revealed the potential interest of STS in the treatment of uremic induced vascular or soft tissues calcifications. Recently, our group has developed an expertise in the use of STS for the treatment of ectopic soft tissue calcifications or ossifications. Considering these promising preliminary data, and their limits, we developed a strategy to treat soft tissue calcifications or ossifications based on a local administration of STS. The first results of this therapeutic strategy are highly promising and the local or systemic safety is satisfactory so far. These preliminary data also reported by others deserve to be confirmed in a prospective study.

We propose in this project to conduct a prospective open controlled phase II trial in order to assess the efficacy and the safety of intralesional administration of STS for the treatment of calcifications secondary to dermatomyositis or systemic sclerosis and ectopic ossifications secondary to pseudo-hypoparathyroidism 1a type (PHP1A/iPPSD2) (inactivating parathyroid hormone / parathyroid-hormone-related peptid (PTH/PTHrP) signalling disorder).

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with:

  * ectopic ossification secondary to iPPSD2 or
  * ectopic calcification secondary to dermatomyositis or
  * ectopic calcification secondary to systemic sclerosis
* Patient aged 2 years or over
* Indication of STS infusion validated by a multidisciplinary committee, based on the significant morbidity and/or functional impact of the targeted calcification/ossification
* Patient with no planned surgery of the calcifications/ossifications for the twelve coming months
* Women of childbearing potential on highly effective contraception (such as hormonal contraception, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner or sexual abstinence)
* Men with women of childbearing potential partners should use condoms during the whole treatment period and until 91 days after the last injection.
* Informed consent signed by the patient / parents
* Patient affiliated to the social security system

Exclusion Criteria:

* Allergy to STS or one of the excipients used
* Contraindication to local injection of STS
* Anticoagulant therapy
* Pregnant, parturient or breastfeeding woman
* Patient deprived of freedom by a court judgment or an administrative decision
* Patient undergoing psychiatric care under coercion
* Legally protected adult patients (guardianship / curatorship)
* Patient unable to give consent
* Patient placed under judicial protection

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2027-06-06 (Estimated); Study Completion 2027-06-06 (Estimated)

PRIMARY OUTCOMES:
Change of the percentage of volume of the treated calcifications / ossifications | between Month 6 and Month 12
  Calculation of percentage of volume evolution of the treated calcification / ossification between the beginning and the end of STS treatment, in each of the three diseases (dermatomyositis, systemic sclerosis and iPPSD2), evaluated on CT-scan measurements.

SECONDARY OUTCOMES:
Change of the volume of the treated calcifications / ossifications | Month 0, Month 6 and Month 12
  Calculation of volume of the treated calcification / ossification at (i) inclusion, the end of the run-in period (6 month) and after 6 months of local injections of STS in each disease (12 month), evaluated on CT-scan measurements.
Adverse events | Month 12
  Collection of adverse events (clinical and biological): causality, severity, and seriousness during the STS treatment.
Change of the Hounsfield density of the treated ectopic calcifications/ossifications | Month 0, Month 6 and Month 12
  Hounsfield density analysis of the treated ectopic calcifications/ossifications at inclusion, the end of the run-in period (6 month) and after 6 months of local injections of STS (12 month), evaluated on CT-scan measurements.
Change of the percentage of patient with a clinically pertinent variation in pain | Between Month0 and Month 6 and Between Month 6 and Month 12
  Calculation of Percentage of patients with a clinically pertinent variation in pain evaluated with pain scales: difference in hetero-evaluation scale of pain in children (HEDEN) ≥ 2 (2-7 years old) between M0-M6 and M6-M12
Change of the percentage of patient with a clinically pertinent variation in pain | Between Month0 and Month 6 and Between Month 6 and Month 12
  Calculation of Percentage of patients with a clinically pertinent variation in pain evaluated with pain scales: difference in visual analogue pain intensity scale (VAS) score ≥ 2 (> 7 years old) between M0-M6 and M6-M12
Change of the percentage of patients with a clinically pertinent variation in quality of life | Between Month0 and Month 6 and Between Month 6 and Month 12
  Calculation of percentage of patients with a clinically pertinent variation in quality of life : difference in PedsQL ≥ 5 (2-18 years old, using appropriates reports) between M0-M6 and M6-M12
Change of the percentage of patients with a clinically pertinent variation in quality of life | Between Month0 and Month 6 and Between Month 6 and Month 12
  Calculation of percentage of patients with a clinically pertinent variation in quality of life : difference in Short Form 36 (SF36) score ≥ 20 (> 18 years old) between M0-M6 and M6-M12

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GUIGONIS, MD, Principal Investigator — University Hospital, Limoges
Locations (8):
- France (8):
  - CHU de BORDEAUX, Bordeaux
  - Hospice Civil de Lyon, Bron
  - ApHp - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU de Limoges, Limoges
  - ApHp - hôpital Lariboisière, Paris
  - Hôpital de la Pitié Salpétriêre, Paris
  - CHU de ROUEN, Rouen
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No